CLINICAL TRIAL: NCT04741724
Title: Effect of Transcutaneous Electrical Diaphragmatic Stimulation in Prolonged Mechanical Ventilation
Brief Title: TEDS in Prolonged Mechanical Ventilation
Acronym: TEDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Chen Yen-Huey, Associate lecture, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201700096A3
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Mechanical Ventilation
Keywords: electrical stimulation; diaphragmatic; weaning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transcutaneous electrical diaphragmatic stimulation (TEDS) (Experimental): Subjects received daily TEDS (30min/day, 5days/week ) until the end of the weaning trial.
  During TEDS, rectangular electrodes were placed on the parasternal region beside the xiphoid process; the sixth and seventh intercostal spaces in line with the mid-axillary line. TEDS was performed by applying biphasic waves at a stimulation frequency of 30 Hz, pulse width of 400 μs. TEDS intensity was gradually increased until visible muscle contraction was observed. Each session lasts for 30 min day.
  Interventions: Device: TEDS
- Control group (No Intervention): Subjects in the control group did not received TEDS program. Subjects in the control group received the same pre- and post-measurement as those in TEDS group. The control group received medical treatment as those in TEDS group. The pulmonary function was measured at the beginning and end of the intervention.

INTERVENTIONS:
Device: TEDS — An non-invasive intervention. During the intervention, the electrode was placed on the skin stimulated muscle.
  Other Names: transcutaneous electrical diaphragmatic stimulation
  Arms: transcutaneous electrical diaphragmatic stimulation (TEDS)

SUMMARY:
Muscle atrophy and diaphragm dysfunction are common with prolonged mechanical ventilation (PMV). Electrical stimulation has been shown to be beneficial in severe chronic heart failure and chronic obstructive pulmonary disease. However, its effect on PMV is unclear. This study examined the effects of transcutaneous electrical diaphragmatic stimulation (TEDS) on respiratory muscle strength and weaning outcomes in patients with PMV.

DETAILED DESCRIPTION:
Subjects on ventilation for ≥21 days were randomly assigned to TEDS or control groups. The TEDS group received muscle electrical stimulation for 30 min/session/day throughout the intervention. Weaning parameters and respiratory muscle strength (Pimax, Pemax) were assessed. The hospitalization outcome, including weaning rate and length of stay, was followed up until discharge.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 20 years;
2. MV for > 6 h/day for > 21 days;
3. medical stability

Exclusion Criteria:

1. acute lung or systemic infection,
2. hemodynamic instability,
3. abdominal distention,
4. pregnancy.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
breathing frequency | through study completion, an average of 2 weeks
  The pulmonary function as assessed by the measurement of respiratory rate
Pimax | through study completion, an average of 2 weeks
  The pulmonary function as assessed by the measurement of max inspiratory pressure
Vt | through study completion, an average of 2 weeks
  The pulmonary function as assessed by the measurement of tidal volume

SECONDARY OUTCOMES:
RCC days | through study completion, an average of 6 weeks
  The total days that participants stay in the respiratory care center
weaning rate | through study completion, an average of 6 weeks
  the status of ventilator use

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Huey Chen, PhD, Study Director — Chang Gung University
Locations (1):
- Dept of Respiratory therapy, Chang Gung University, Taoyuan District, Taiwan